CLINICAL TRIAL: NCT07250672
Title: Examining the Effect of Action Observation Training Using Patient-Specific 3D Records in Parkinson's Patients
Brief Title: Patient-Specific 3D Action Observation Training in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, enes tayyip benli, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-BENLI-009
Record Dates: First submitted 2025-10-02; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Virtual Reality; Action Obervation Training; Immersive Virtual Reality; 3d Recording
Keywords: Parkinson; Virtual reality
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study will use a randomized, parallel-group, interventional design.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-Specific VR Group (Experimental): Participants will undergo action observation training delivered in immersive virtual reality using their own 3D motion recordings.
  Interventions: Other: Patient-Specific VR Action Observation Training
- Healthy-Model VR Group (Active Comparator): Participants will undergo action observation training delivered in immersive virtual reality using 3D recordings obtained from healthy individuals performing the same actions.
  Interventions: Other: Healthy-Model VR Action Observation Training

INTERVENTIONS:
Other: Patient-Specific VR Action Observation Training — Participants will receive immersive VR action observation training using their own 3D motion recordings captured with an Insta360 camera (Arashi Vision Inc., Shenzhen, China). In Parkinson's patients, only the initial movement sequences without bradykinetic slowing will be selected, and these will be extended to the desired duration using loop playback or ping-pong loop playback in the device's proprietary software. The action observation protocol will consist of the following one-minute tasks: (1) total finger abduction and adduction, (2) fist making and opening, (3) wrist flexion and extension, (4) forearm pronation and supination, and (5) rhythmic striking of the dorsal and palmar surfaces of one hand against the palm of the other. A 1-minute rest will be given between each video. Training will be provided in addition to conventional therapy (35 minutes, 3 days per week for 6 weeks) tailored to individual needs.
  Arms: Patient-Specific VR Group
Other: Healthy-Model VR Action Observation Training — Participants will receive immersive VR action observation training using 3D video recordings of the same activities performed by healthy individuals, captured with an Insta360 camera (Arashi Vision Inc., Shenzhen, China). Recordings will not require editing or adjustments. The action observation protocol will consist of the same one-minute tasks: (1) total finger abduction and adduction, (2) fist making and opening, (3) wrist flexion and extension, (4) forearm pronation and supination, and (5) rhythmic striking of the dorsal and palmar surfaces of one hand against the palm of the other. A 1-minute rest will be given between each video. Training will be provided in addition to conventional therapy (35 minutes, 3 days per week for 6 weeks) tailored to individual needs.
  Arms: Healthy-Model VR Group

SUMMARY:
Although studies exist demonstrating the effects of single-session action observation training on bradykinesia in patients with Parkinson's disease, research investigating the long-term application of such training remains limited. Furthermore, the broader literature indicates that action observation training has typically been conducted in simulated environments or by using recordings obtained from healthy individuals. The aim of the present study is to examine the effects of action observation training, delivered in a fully immersive virtual reality environment using each patient's own 3D motion recordings, on bradykinesia and other disease-related parameters.

DETAILED DESCRIPTION:
Action observation training has been applied across diverse populations to improve performance and treat pathological conditions. Considering that bradykinesia tends to manifest more prominently in rhythmic movements, studies in healthy individuals have shown that merely observing rhythmic actions can influence spontaneous finger movement speed and lead to changes in motor performance, thereby paving the way for the use of action observation in addressing bradykinesia. In a study investigating the effects of action observation in patients with Parkinson's disease, observing fast rhythmic finger movements was reported to increase spontaneous finger movement speed, and compared with acoustic training, the effect of action observation persisted longer over time. Research on imagery through action observation further indicates that immersive virtual reality headsets, compared to monitor screens, facilitate the development of more distinct spatial rhythmic patterns in the brain. This evidence supports the use of fully immersive VR headsets instead of non-immersive monitor-based systems in action observation training.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to participate in the study
* Clinical diagnosis of Parkinson's disease confirmed by a neurologist
* Ongoing treatment with antiparkinsonian medication
* Hoehn and Yahr (H-Y) stage ≤ 3
* Ability to walk independently

Exclusion Criteria:

* Presence of additional neurological disorders other than Parkinson's disease
* Change in medication dosage within the past month
* Score of ≥ 10 on the Simulator Sickness Questionnaire
* Presence of amblyopia, strabismus, or pathologies impairing focus, depth perception, or normal 3D vision
* Failure on the butterfly test of the Titmus stereotest (greater than 3,552 seconds of arc)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Movement Rate (SMR | At baseline and after completion of 6-week intervention period
  In this study, kinematic parameters of finger movements will be determined from video recordings. A commercial motion analysis software will be used to extract the coordinates of manually marked tracking points, which will then be transferred into tabular form for analysis. To improve the accuracy of marking and tracking, participants will wear fingertip gloves in different colors.The spontaneous movement rate will be calculated from video-recorded finger-tapping tasks. Each cycle consists of a touch duration (TD) and an inter-tapping interval (ITI). SMR will be defined as the inverse of the total duration of one tapping cycle (TD + ITI) and expressed in Hertz (Hz).

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | At baseline and after completion of 6-week intervention period
  Disease severity will be assessed using the Unified Parkinson's Disease Rating Scale (UPDRS), the most commonly used valid and reliable instrument for evaluating impairments and disabilities in Parkinson's disease.
Nine-Hole Peg Test (NHPT) | At baseline and after completion of 6-week intervention period
  The Nine-Hole Peg Test is a performance-based assessment of manual dexterity. Before the test begins, participants will be instructed and shown how to perform the task once. They will then be asked to pick up the pegs one by one, place them into the holes, and after filling all holes, remove them one by one and place them back into the container.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | At baseline and after completion of 6-week intervention period
  The Disabilities of the Arm, Shoulder and Hand Questionnaire is a 30-item instrument used to evaluate upper extremity function and the impact of upper limb problems on daily activities. The first 21 items assess the degree of difficulty in performing various daily activities with the dominant extremity over the past week. The next 5 items assess the severity of pain, numbness, and weakness experienced during activities. The final 4 items evaluate the impact of upper limb pathology on sleep, work, social life, and psychological status.
Parkinson's Disease Questionnaire (PDQ-8) | At baseline and after completion of 6-week intervention period
  Quality of life in Parkinson's disease will be assessed using the Parkinson's Disease Questionnaire (PDQ-39), a disease-specific instrument consisting of 39 items across eight domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (3 items), social support (3 items), cognition (4 items), communication (3 items), and bodily discomfort (4 items). To reduce participant burden, the PDQ-8, a short form including one representative item from each domain, may also be used. Items in the PDQ-8 evaluate the patient's status over the past month and are scored on a 5-point scale ranging from 0 (never) to 4 (always).
Intrinsic Motivation Inventory (IMI) | After completion of 6-week intervention period
  The Intrinsic Motivation Inventory (IMI) is a multidimensional questionnaire used to assess participants' motivation and satisfaction while performing a given activity. It evaluates several domains, including interest/enjoyment, perceived competence, pressure/tension, perceived choice, and value/usefulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, individual participant data (IPD) will not be made available to other researchers.